CLINICAL TRIAL: NCT06336395
Title: Ma-Spore ALL-Seq 2020: RNA-Seq and IgH/TCR-Seq to Improve Risk Assignment in Childhood, Adolescent and Young Adult Acute Lymphoblastic Leukaemia
Brief Title: Ma-Spore ALL 2020 Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/00888
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: B Lymphoblastic Leukemia
MeSH Terms: interventions — Prednisolone; Dexamethasone; Vincristine; Methotrexate; Asparaginase; pegaspargase; Dasatinib; Imatinib Mesylate; Cyclophosphamide; Cytarabine; Mercaptopurine; Thioguanine; Rituximab; Doxorubicin; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard risk (SR) (Experimental): 1. No anthracycline throughout the treatment.
  2. CNS consolidation using "Capizzi type" low dose methotrexate (LDMTX) x 2 courses to replace pre-existing high dose methotrexate (HDMTX) 2.5g #3/4
  Interventions: Drug: Prednisolone; Drug: Dexamethasone; Drug: Vincristine; Drug: Methotrexate; Drug: L-Asparaginase; Drug: Pegylated asparaginase; Drug: Erwinase; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Mercaptopurine; Drug: Thioguanine
- Intermediate risk (IR) (Experimental): Those with CD20 ≥ 20% expression on diagnostic blasts by flow immunophenotyping will receive additional dose of rituximab on day 1 of each delayed intensification (DI) phases: phase III (2 courses) and V (1 course) for total 3 infusions
  Interventions: Drug: Prednisolone; Drug: Dexamethasone; Drug: Vincristine; Drug: Methotrexate; Drug: L-Asparaginase; Drug: Pegylated asparaginase; Drug: Erwinase; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Mercaptopurine; Drug: Thioguanine; Drug: Rituximab; Drug: Doxorubicin
- High risk (HR) (Experimental): Provisional HR patients will be offered CAR-T cell immunotherapy or HSCT
  Interventions: Drug: Prednisolone; Drug: Dexamethasone; Drug: Vincristine; Drug: Methotrexate; Drug: L-Asparaginase; Drug: Pegylated asparaginase; Drug: Erwinase; Drug: Dasatinib; Drug: Imatinib; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Mercaptopurine; Drug: Thioguanine; Drug: Doxorubicin; Drug: Fludarabine

INTERVENTIONS:
Drug: Prednisolone — Oral
Drug: Dexamethasone — Oral
Drug: Vincristine — Intravenous
Drug: Methotrexate — Oral/ intrathecal/intravenous/subcutaneous
Drug: L-Asparaginase — Intramuscular
Drug: Pegylated asparaginase — Intravenous
Drug: Erwinase — Optional for those allergic to E.coli/PEG L-asparaginase (intravenous)
Drug: Dasatinib — Indicated only for ALL with BCR::ABL1 /BCR::ABL1-like/ tyrosine kinase fusion positive (oral)
  Arms: High risk (HR)
Drug: Imatinib — Indicated only for ALL with BCR::ABL1 /BCR::ABL1-like/ tyrosine kinase fusion positive (oral)
  Arms: High risk (HR)
Drug: Cyclophosphamide — Intravenous
Drug: Cytarabine — Subcutaneous/ Intravenous
Drug: Mercaptopurine — Oral
Drug: Thioguanine — Oral
Drug: Rituximab — Intravenous
  Arms: Intermediate risk (IR)
Drug: Doxorubicin — Intravenous
  Arms: High risk (HR); Intermediate risk (IR)
Drug: Fludarabine — Intravenous
  Arms: High risk (HR)

SUMMARY:
The primary objective of this trial is to improve the overall survival rate of children and young adult with B-lineage acute lymphoblastic leukemia (B-ALL) in Singapore and Malaysia in the context of a multicenter cooperative trial using a risk-stratified therapy.

DETAILED DESCRIPTION:
This is a multicenter open-label phase II study involving children and young adult (< 41 years old) who are newly diagnosed with B-ALL and treatment naïve. There will be 3 parallel cohorts whose risk to be stratified based upon leukemia genetics profiles and patient's treatment response:

1. Standard Risk (SR)
2. Intermediate Risk (IR)
3. High Risk (HR)

All drugs being used are commercially available chemotherapy drugs. There will be no novel chemotherapeutic agent without marketing authorization being tested in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Has been diagnosed with B-lineage ALL as evidenced by:

   1. BMA blasts > 20% AND
   2. Leukemic process in the bone marrow, peripheral blood or any extra medullary tissue with confirmation of B-lymphoid differentiation by flow immunophenotyping or histopathologically
2. Age < 41 years of age at enrolment
3. Written informed consent obtained from patient or legally acceptable representative (LAR)

Exclusion Criteria:

1. T-lineage ALL
2. Down syndrome with ALL
3. History of previous malignancies or this ALL is a second malignancy
4. Mixed phenotype acute leukemia (MPAL) or undifferentiated leukemia
5. Mature B-cell leukemia/lymphoma
6. Any previous cytotoxic therapy (chemotherapy/radiotherapy/immunotherapy). Patient pre-treated with short term steroid (< 7 days of duration within last 1 month prior to ALL treatment start) may be enrolled after discussion and written approval from PI. These patients should be treated on at least intermediate arm.
7. Persistent renal dysfunction with creatinine more than upper limit of normal for age before start of induction therapy. Patients requiring temporary dialysis without persistent renal dysfunction can qualify.
8. Liver dysfunction with direct bilirubin > 10x upper normal limit for age.
9. Any serious uncontrolled medical condition or impending end organ dysfunction that would impair the ability of the subject to receive protocol therapy
10. Doubtful compliance or ability to complete study therapy due to financial, social, familial or geographic reason, or in the judgement of site investigator

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-03-04 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 5 years from diagnosis
  OS is calculated from the date of diagnosis to the date of last follow-up or any death

SECONDARY OUTCOMES:
Event free survival (EFS) | 5 years from diagnosis
  EFS will be calculated from the date of diagnosis of ALL to date of last follow-up or to the first event, including relapse, resistant disease, second malignancy and death

OTHER OUTCOMES:
Cumulative incidence (CI) of relapse for all treated cohorts | 5 years from diagnosis
Cumulative incidence (CI) of therapy-related mortality (TRM) for all treated subjects | 5 years from diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Allen Eng Juh Yeoh, MBBS, Principal Investigator — Professor
Locations (3):
- Malaysia (2):
  - Subang Jaya Medical Centre, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No